CLINICAL TRIAL: NCT01091584
Title: A Randomized Trial to Assess the (Cost) Effectiveness of the Use of the Distress Thermometer by a Nurse in Addition to Usual Care for Patients Treated With Curative Intent for Breast Cancer.
Brief Title: Nurse Intervention Project
Acronym: VIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CMO: 2009/293
Record Dates: First submitted 2010-03-17; First posted 2010-03-24 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-11

CONDITIONS: Breast Cancer Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- intervention group (Active Comparator): The intervention is to apply the distress thermometer as written in the guideline written by 'Vereniging Integrale Kankercentra' title: 'Detecteren behoefte psychosociale zorg. The distress thermometer is collected from the experimental group and then discussed by a trained nurse.
  Interventions: Device: distress thermometer
- control group (No Intervention): usual care

INTERVENTIONS:
Device: distress thermometer — to apply the distress thermometer as written in the guideline written by 'Vereniging Integrale Kankercentra' title: 'Detecteren behoefte psychosociale zorg. The distress thermometer is collected from the experimental group and then discussed by a trained nurse
  Arms: intervention group

SUMMARY:
The use of interventions for cancer-related distress is important to reduce this distress. Distress has a negative impact on quality of life, the recovery during and after treatment and may even adversely affect survival. There is insufficient attention to the systematic approach to psychosocial problems in cancer patients in the Netherlands. A task force discussed and studied which instrument measures psychosocial problems best. The distress thermometer ("lastmeter") had the best results. A guideline is written to use the distress thermometer for patients with cancer and will be used in hospitals in the Netherlands. However, it is not clear what the effects are of the use of the distress thermometer on the psychosocial wellbeing of the patient. Furthermore, it is also unknown whether the use of the distress thermometer leads to cost-effective care. The study focuses on the use of the distress thermometer in breast cancer patients. An efficiency study (RCT) will be conducted to evaluate the systematic use of the distress thermometer and its discussion by a nurse as compared to the usual care provided to outpatients who are treated with curative intent for breast cancer by their treating physicians. The clinical and economic impact of the use of the Distress thermometer will be assessed in comparison with usual care.The recruitment of patients will take place in the out-patient clinic of a university hospital. Patients will be followed from diagnose until two years after finishing their treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven malignancy of the breast
* Curative treatment
* Dominated the dutch language
* Age > 18 year

Exclusion Criteria:

* Previously treated for a malignancy
* Psychiatric problems that adherence this study

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2010-03; Primary Completion 2013-02 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Subscale quality of life of the questionnaire: EORTC QLQ C30 | After each treatment completion, during follow up; first year every 3 months, second year every 6 months
  Subscale quality of life of the questionnaire: EORTC QLQ C30

SECONDARY OUTCOMES:
Other subscales | After each treatment completion, during follow up; first year every 3 months, second year every 6 months
  Other subscales:
  * HADS : anxiety and depression
  * EORTC BR23 : breast cancer specific problems
  * SVL: Impact of Event Scale
  * ZCL : illness cognition questionnaire with subscales: disease benefits, acceptance and helplessness
  * EuroQoL6D,
  * Cost diary

CONTACTS AND LOCATIONS:
Overall Officials: P. B. Ottevanger, Dr, Principal Investigator — University Medical Centre Nijmegen
Locations (1):
- University Medical Centre Nijmegen, Nijmegen, Netherlands

REFERENCES:
- [Derived] Ploos van Amstel FK, Prins JB, van der Graaf WT, Peters ME, Ottevanger PB. The effectiveness of a nurse-led intervention with the distress thermometer for patients treated with curative intent for breast cancer: design of a randomized controlled trial. BMC Cancer. 2016 Jul 25;16:520. doi: 10.1186/s12885-016-2565-x. PMID 27455960